CLINICAL TRIAL: NCT04770480
Title: Exploring Non-pharmacological Approaches to Pain Management After Lumbar Surgery: A Randomized Controlled Trial
Brief Title: Non-pharmacological Treatment for Pain After Spine Surgery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dan Rhon (U.S. Federal Agency)
Collaborators: University of Utah (Other); Madigan Army Medical Center (U.S. Federal Agency); Tripler Army Medical Center (U.S. Federal Agency); 59th Medical Wing (U.S. Federal Agency); National Center for Complementary and Integrative Health (NCCIH) (NIH); Brooke Army Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Dan Rhon, Director, Primary Care Musculoskeletal Research Center, Brooke Army Medical Center
Organization: Brooke Army Medical Center (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: eIRB; 3UH3AT009763-04S1 (NIH)
Record Dates: First submitted 2021-02-22; First posted 2021-02-25 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Low Back Pain; Chronic Pain; Surgery; Back Pain, Low; Back Pain Lower Back Chronic
Keywords: chronic pain; low back pain; spine surgery; non-pharmacological treatment; mindfulness; physical therapy
MeSH Terms: conditions — Low Back Pain; Chronic Pain | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Primary Outcome: The primary analysis will be performed by fitting a longitudinal linear model to the PEG scores at baseline, 2 weeks and 26 weeks.
  Secondary Outcome: Kaplan Meier curves with 95% pointwise confidence limits will be constructed to summarize the time to opioid discontinuation in each of the EPM and SC treatment groups. Time to opioid discontinuation will be compared between groups using a stratified log-rank test, with stratification for three randomization stratification factors.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Study participants and clinicians cannot be blinded to study treatments. Randomization assignment will not be revealed until after enrollment and completion of baseline assessments. Study statisticians cannot be blinded to participants' study treatment assignments because they must complete Data Safety Monitoring Reports and analyze the study outcomes by treatment group. Study investigators will remain blinded to participants' treatment group assignment. Follow-up assessments will be performed by a research assistant who will be blinded to participants' treatment group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care (SC) (Active Comparator): Standard Post-Surgical Care utilizing opioids.
  Interventions: Behavioral: Standard Care (SC)
- Enriched Surgical Management Pathway (EMP) (Active Comparator): Enriched Surgical Management Pathway utilizing Physical Therapy and Mindfulness in addition to Standard Protocol.
  Interventions: Behavioral: Enriched Pain Management Pathway (EPM)

INTERVENTIONS:
Behavioral: Standard Care (SC) — No attempt will be made to change usual care practice after surgery
  Arms: Standard Care (SC)
Behavioral: Enriched Pain Management Pathway (EPM) — Enriched Pain Management Pathway will be delivered by physical therapists trained to integrate physical therapy and mindfulness techniques grounded in a biopsychosocial context. The intervention will be delivered within the context of the post-operative physical therapy routine (the mindfulness approach will be integrated into the post-operative physical therapy care).
  Arms: Enriched Surgical Management Pathway (EMP)

SUMMARY:
This study will compare the effectiveness of two pain management pathways (standard vs. enriched) for patients undergoing lumbar spine surgery in the Military Health System (MHS). Effectiveness will be based on post-surgery patient-centered outcomes and extent of opioid use. The study design is a 2-arm, parallel group, individual-randomized trial.

DETAILED DESCRIPTION:
The relevance of our model is supported by evidence that pain catastrophizing, self-efficacy and hypervigilance predict poor surgical outcomes and long-term opioid use. Surgery can exacerbate catastrophic thinking, especially if patients have unrealistic recovery expectations that go unmet. Physical therapy (PT) can improve chronic LBP (low back pain) outcomes, with effects mediated through changes in pain catastrophizing and self-efficacy. Mindfulness techniques help patients disentangle an experience (e.g., pain) from associated emotions and appraisals. Mindfulness can enhance emotion regulation and raise un-conscious behavioral responses (e.g., opioid use) to conscious consideration. The benefits of mindfulness for chronic pain are mediated by changes in hypervigilance and self-efficacy. Physical therapy and mindfulness can disrupt the self-reinforcing cycle of pain, catastrophic appraisal and unconscious behavioral response including opioid use. Our project examines an innovative strategy to integrate mindfulness and PT into an enriched surgical management pathway for individuals undergoing lumbar spine surgery.

Patients at 3 different military hospitals will be randomized prior to surgery to two different treatment groups and followed for a period of 6 months, including the post-operative intervention phase.

ELIGIBILITY:
Inclusion Criteria:

1. Tricare beneficiary receiving care in a participating MHS facility.
2. Age 18 - 75 years at the time of enrollment
3. Scheduled to undergo lumbar spine surgery within the next 60 days. Surgery may be laminectomy with or without fusions including lateral, transforaminal, posterior or anterior approach for 1-4 lumbar levels. Surgery may be performed in military or civilian facility
4. Indication for surgery may include disc herniation, degenerative disc disease, lumbar stenosis, degenerative spondylolisthesis or scoliosis.
5. Anticipates ability to attend treatment sessions over a 16 week period following the surgical procedure with no planned absence of 2 weeks or more for training, vacation or any purpose

Exclusion Criteria:

1. Indication for surgery is infection, fracture, tumor, trauma or other indication requiring emergency surgery.
2. A microsurgical technique as the primary procedure, such as an isolated laminotomy or microdiscectomy
3. Surgical procedure is a revision or participant has undergone a lumbar surgical procedure in the past year.
4. Contra-indication to participation in post-operative exercise program including severe orthopedic injury limiting mobility, wheelchair dependency, neurological disorder impacting mobility, reliance on supplemental oxygen for daily activity, etc.
5. Pending a medical evaluation board, discharge from the military for medical reasons, or pending or undergoing any litigation for an injury

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 267 (Actual)
Dates: Start 2021-12-10 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Pain, Enjoyment, and General Activity Scale (PEG-3) | 6 Months
  The PEG-3 measure includes 3 items evaluating 1) pain severity, and interference of pain with 2) enjoyment and 3) general activity. Response options for each item range from 0-10 with higher scores indicating higher pain intensity. The PEG-3 score is expressed as the mean of all item scores.

SECONDARY OUTCOMES:
Time to Discontinuation of Opioids After Surgery | 6 Months
  The length of time (recorded in days) until a patient discontinues pain medications after surgery.

OTHER OUTCOMES:
Patient-Reported Outcomes Measurement Information System (PROMIS)-29 version 2.0 | 6 months
  The PROMIS-29 measures 7 domains of health-related quality of life (pain interference, physical function, anxiety, depression, sleep disturbance, fatigue, and ability to participate in social roles) using 4 items and includes a single 0-10 numeric pain intensity rating scale. Scores are provided as T-scores for all domains and can be used to compute a mental and physical health summary score

CONTACTS AND LOCATIONS:
Overall Officials: Julie M Fritz, PhD, Principal Investigator — University of Utah; Daniel I Rhon, DSc, Principal Investigator — Brooke Army Medical Center
Locations (3):
- United States (3):
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Brooke Army Medical Center, San Antonio, Texas
  - Madigan Army Medical Center, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: Yes
Trial data from this trial will be entered into the National Institutes of Health Help End Addiction Long-Term (HEAL)Back Pain Consortium (BACPAC) data repository and coordinating center.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Within 6 months of completion of all trial activities.
Access Criteria: Requests to use data from the BACPAC data repository need to go through that organization. Otherwise, reasonable requests will be considered as long as all data sharing agreement (DSA) stipulations from the US Defense Health Agency have been met. More about filling out and submitting DSAs can be found at https://www.health.mil/
URL: https://www.health.mil/Military-Health-Topics/Privacy-and-Civil-Liberties/Submit-a-Data-Sharing-Application

REFERENCES:
- [Background] Deyo RA, Hallvik SE, Hildebran C, Marino M, O'Kane N, Carson J, Van Otterloo J, Wright DA, Millet LM, Wakeland W. Use of prescription opioids before and after an operation for chronic pain (lumbar fusion surgery). Pain. 2018 Jun;159(6):1147-1154. doi: 10.1097/j.pain.0000000000001202. PMID 29521813
- [Background] Weinstein JN, Tosteson TD, Lurie JD, Tosteson AN, Hanscom B, Skinner JS, Abdu WA, Hilibrand AS, Boden SD, Deyo RA. Surgical vs nonoperative treatment for lumbar disk herniation: the Spine Patient Outcomes Research Trial (SPORT): a randomized trial. JAMA. 2006 Nov 22;296(20):2441-50. doi: 10.1001/jama.296.20.2441. PMID 17119140
- [Background] Ong KL, Stoner KE, Yun BM, Lau E, Edidin AA. Baseline and postfusion opioid burden for patients with low back pain. Am J Manag Care. 2018 Aug 1;24(8):e234-e240. PMID 30130023
- [Background] Woby SR, Urmston M, Watson PJ. Self-efficacy mediates the relation between pain-related fear and outcome in chronic low back pain patients. Eur J Pain. 2007 Oct;11(7):711-8. doi: 10.1016/j.ejpain.2006.10.009. Epub 2007 Jan 10. PMID 17218132
- [Background] Morasco BJ, Yarborough BJ, Smith NX, Dobscha SK, Deyo RA, Perrin NA, Green CA. Higher Prescription Opioid Dose is Associated With Worse Patient-Reported Pain Outcomes and More Health Care Utilization. J Pain. 2017 Apr;18(4):437-445. doi: 10.1016/j.jpain.2016.12.004. Epub 2016 Dec 18. PMID 27993558
- [Background] Fritz JM, Magel JS, McFadden M, Asche C, Thackeray A, Meier W, Brennan G. Early Physical Therapy vs Usual Care in Patients With Recent-Onset Low Back Pain: A Randomized Clinical Trial. JAMA. 2015 Oct 13;314(14):1459-67. doi: 10.1001/jama.2015.11648. PMID 26461996
- [Background] Rhon DI, Miller RB, Fritz JM. Effectiveness and Downstream Healthcare Utilization for Patients That Received Early Physical Therapy Versus Usual Care for Low Back Pain: A Randomized Clinical Trial. Spine (Phila Pa 1976). 2018 Oct 1;43(19):1313-1321. doi: 10.1097/BRS.0000000000002619. PMID 29489568
- [Background] Lo YT, Lim-Watson M, Seo Y, Fluetsch N, Alasmari MM, Alsheikh MY, Lamba N, Smith TR, Aglio LS, Mekary RA. Long-Term Opioid Prescriptions After Spine Surgery: A Meta-Analysis of Prevalence and Risk Factors. World Neurosurg. 2020 Sep;141:e894-e920. doi: 10.1016/j.wneu.2020.06.081. Epub 2020 Jun 19. PMID 32569762
- [Background] Siglin J, Sorkin JD, Namiranian K. Incidence of Postoperative Opioid Overdose and New Diagnosis of Opioid Use Disorder Among US Veterans. Am J Addict. 2020 Jul;29(4):295-304. doi: 10.1111/ajad.13022. Epub 2020 Mar 22. PMID 32202000
- [Background] Schoenfeld AJ, Belmont PJ Jr, Blucher JA, Jiang W, Chaudhary MA, Koehlmoos T, Kang JD, Haider AH. Sustained Preoperative Opioid Use Is a Predictor of Continued Use Following Spine Surgery. J Bone Joint Surg Am. 2018 Jun 6;100(11):914-921. doi: 10.2106/JBJS.17.00862. PMID 29870441
- See also: HEAL BACPAC — https://heal.nih.gov/research/clinical-research/back-pain